CLINICAL TRIAL: NCT00060593
Title: Self-Perception of Postural Stability: Event-Related fMRI Study
Brief Title: MRI Study of Self-Perception of Postural Stability
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030183; 03-N-0183
Record Dates: First submitted 2003-05-07; First posted 2003-05-08 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-05

CONDITIONS: Healthy; Postural Stability
Keywords: Balance; Functional Connectivity; Healthy Volunteer; HV

SUMMARY:
This study will use functional magnetic resonance imaging (MRI) to examine loss of balance in the elderly. Falls due to balance problems are a major health issue in older people, often resulting in bone fractures and other bodily injuries, and in functional decline. Risk factors for falling in the elderly include some standing positions in which older people usually experience balance problems, such as leaning forwards or backwards. Functional MRI records brain function while the subject performs a task, such as moving a limb or speaking, and detects changes in the brain regions involved in those tasks. This study will look at different brain areas to see which areas might control what people see around them while they are standing.

Healthy normal volunteers between 20 and 90 years of age may be eligible for this study. Candidates must be in good health, have no difficulties in performing activities of daily living, and be able to walk for at least 400 meters (1/4 mile). They will be screened with a medical history and physical examination.

Participants will undergo functional MRI while performing visual recognition tasks in two experiments, described below. For the MRI procedure, the subject lies in the MRI scanner, a narrow metal cylinder containing a strong magnet, for 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. The experiments are as follows:

Experiment 1

During MRI scanning, the subject watches computer-generated movies of a person leaning forwards and backwards. When the subject recognizes an unstable body position in the movements, he or she presses a computer mouse.

Experiment 2

During MRI scanning, the subject watches still pictures of people leaning in stable and unstable postures and presses a button as soon as he or she recognizes that the posture is unstable.

DETAILED DESCRIPTION:
A number of studies have explored the role of visual, vestibular and somatosensory systems in the control of upright posture. However, the cortical control of postural stability, in general, and the role of higher cognitive function in assessment of postural stability, in specific, has not been studied extensively. It is well established that certain features of postural control change during the advancing years of life so that the stability of posture can be a problem in the elderly. However, neural mechanisms of postural stability that decline with age and make older adults more prone to falling have not been identified specifically. To characterize specific causes of falling in the elderly is problematic, because human posture is a product of an extremely complex dynamical system and like any other physical activity undergoes dramatic changes in organization throughout the life-span. In our previous research we showed the neural activation patterns embodied in the electroencephalogram (EEG) were associated with recognition of unstable postures in young healthy subjects. In another protocol, we propose that these patterns will systematically change with aging, and will result in difficulty to discriminate relevant from irrelevant information in the control of upright posture. The present study focuses on the evaluation of neural activation patterns underlying recognition of unstable postures in 15 young controls and 15 elderly subjects using both the block and event-related functional MRI (fMRI) designs. We will first analyze how the frontal-parieto-occipital circuits play a role in perception of postural stability in young subjects and then perform similar studies using elderly subjects. After the fMRI measurements a detailed evaluation of the haemodynamic response (BOLD) signals will be performed. Further analysis will look at the functional connectivity between the motion-selective cortical area (V5), the posterior parietal cortex (PP) and the frontal cortex (FC), using correlation methods. It is expected that from the study will uncover important insights in neural mechanisms as it relates to the self-perception of postural stability and its deterioration as a result of aging.

ELIGIBILITY:
INCLUSION CRITERIA:

There will be 20 subjects in each aforementioned age group.

Subjects will be enrolled in this study if they are within the range of 20-50 (young group) and 70-90 (old group) years old, in good health, report no difficulties or need for help in performing self-care or instrumental activities of daily living, are able to walk for at least 400 meters.

All subjects and patients participating in this study will have a valid Clinical Center Medical Record Number.

EXCLUSION CRITERIA:

We will be unable to study people who have substantial cognitive impairment based on mental status screening tests, history of cardiovascular disease (including angina, myocardial infarction, congestive heart failure, cerebro-vascular disease), cancer, neurological diseases, birth defects, kidney or liver disease, gastrointestinal (G.I.) disease, musculo-skeletal disorder (if they cause pathological weakness and/or chronic pain), important sensory deficits and any conditions that precludes them from being tested with standard neuropsychological tests.

MRI experiments will not be performed in subjects or patients who have pacemakers, brain stimulators, dental implants or metallic braces, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, insulin pump, or shrapnel fragments.

We will not scan pregnant women because of the safety of high magnetic fields to the fetus is not established.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-05; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Arfken CL, Lach HW, Birge SJ, Miller JP. The prevalence and correlates of fear of falling in elderly persons living in the community. Am J Public Health. 1994 Apr;84(4):565-70. doi: 10.2105/ajph.84.4.565. PMID 8154557
- [Background] Bandettini PA, Jesmanowicz A, Wong EC, Hyde JS. Processing strategies for time-course data sets in functional MRI of the human brain. Magn Reson Med. 1993 Aug;30(2):161-73. doi: 10.1002/mrm.1910300204. PMID 8366797
- [Background] Basar E, Demiralp T. Fast rhythms in the hippocampus are a part of the diffuse gamma-response system. Hippocampus. 1995;5(3):240-1. doi: 10.1002/hipo.450050311. No abstract available. PMID 7550619